CLINICAL TRIAL: NCT04672720
Title: The Effect of Adding L-carnitine During Ovarian Stimulation With Antagonistic Protocol in Patients With Polycystic Ovarian Syndrome on the Outcome of IVF / ICSI Cycle: A Double Blind Randomized Clinical Trial
Brief Title: L-carnitine and COH in PCOS Women Undergoing IVF/ICSI Cycles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: L-carnitine - PCOS- ART
Record Dates: First submitted 2020-12-13; First posted 2020-12-17 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Polycystic Ovary Syndrome
Keywords: L-carnitine; Assisted reproductive technology; Controlled ovarian stimulation
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Carnitine; Quaternary Ammonium Compounds

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: L-carnitine and placebo drugs can be identified only by special codes determined by a statistics specialist. The participant, care provider, investigator and outcome assessor are unaware of the type of study groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adding l-carnitine to controlled ovarian stimulation antagonist protocol (Experimental): The controlled ovarian stimulation procedure in all the study participate will be same by using a flexible regimen of GnRH antagonist with E2 priming. In the experimental group, the women will receive 3 tablet of L-carnitine daily (L-carnitine® tablet 1000 mg, Karen Pharmaceutical Company, Iran) from day 2 of the previous menstrual cycle until pregnancy test day.
  Interventions: Drug: L-carnitine 1000 Mg
- Adding placebo to controlled ovarian stimulation antagonist protocol (Placebo Comparator): The controlled ovarian stimulation procedure in all the study participate will be same by using a flexible regimen of GnRH antagonist with E2 priming. The patients in the control group will receive 3 placebo tablets in similar way for 8 weeks.
  Interventions: Drug: L-carnitine 1000 Mg

INTERVENTIONS:
Drug: L-carnitine 1000 Mg — Prescription 3mg l-carnitine (L-carnitine® tablet 1000 mg, Karen Pharmaceutical Company, Iran) daily from day 2 of the previous menstrual cycle until pregnancy test day (approximately 8 weeks).
  Other Names: Quaternary ammonium compound

SUMMARY:
The aim of this study was to evaluate the effect of oral L-carnitine supplementation during controlled ovarian stimulation (COS) in patients with polycystic ovary syndrome (PCOS) in a double-blind randomized clinical trial. The eligible patients with PCOS diagnosis (on the basis of Rotterdam criteria) who referred to Royan Research Institute for IVF / ICSI treatment cycles will be evaluated.

DETAILED DESCRIPTION:
The study protocol was approved by the Institutional Review Board and Ethics Committee of Royan institute. Prior to the onset of ovarian stimulation, patients will be allocated randomly into two groups according to block randomization method. The methodologist will give the doctor a code according to the randomization list, which corresponds to the code on the drug's box, and the drug box will be delivered to the patient. The COS procedure in all the study participate will be same by using a flexible regimen of GnRH antagonist with E2 priming. In the experimental group, the women received 3 tablet of L-carnitine daily (L-carnitine® tablet 1000 mg, Karen Pharmaceutical Company, Iran) from day 2 of the previous menstrual cycle until pregnancy test day. The patients in control group will receive 3 placebo tablets for 8 weeks. All the placebo tablets were produced by Karen company (Tehran, Iran), which is approved by the Food and Drug Administration of Iran. The appearance of the placebo was indistinguishable in color, shape, size, and smell from L-carnitine tablets. Ovarian stimulation will start with a maximum dose of 150 units of rFSH (Gonal -F: Serono Laboratories Ltd, Geneva, Switzerlan), from the second or third day of the spontaneous or discontinued progesterone menstrual cycle and the monitoring transvaginal ultrasound was performed and then if the follicle is observed, start with 13 injections of GnRH antagonist (Cetrotide®, 0.25 mg cetrorelix acetate, Serono, Inc) and will be continued until the oocyte triggering day. From the seventh day of the cycle, the dose of rFSH will be determined according to the rate of ovarian response by vaginal ultrasonography two days in advance. If you see at least two follicles 18 mm in size or more, the final stimulation of oocyte maturation will be done and 34- 36 hour after that the ovum pickup will be conducted. Subsequently ICSI or IVF will be done with standard procedure. In the present study, the markers of insulin metabolism (fasting glucose and insulin) and lipid profiles (LDL, HDL, cholesterol and triglyceride) as well as body mass index and weight were measured at the baseline of the study (before starting L-carnitine supplementation) as well as 6 weeks later on the ovum pick up day.The outcome evaluators were also blinded to the random allocation process and type of treatment.The primary and secondary outcomes were compared between the two groups using appropriate statistical tests.

ELIGIBILITY:
Inclusion Criteria:

• Patients between 20 to 37 years old, presenting with primary or secondary infertility following regular intercourse for at least 1 year and diagnosed with polycystic ovary syndrome (PCOS) according to Rotterdam's criteria who had received two to three failures of IUI cycle therapy were included. The diagnosis was based on a complete history taking, physical examination and a paper documented complete infertility work-up within the previous 6 months

Exclusion Criteria:

1. Patients diagnosed with hyperprolactinemia, diabetes mellitus, epilepsy
2. Patients treated with special diet, medication supplement (ovuboost), metformin before or during ovarian stimulation
3. History of pelvic surgery on ovaries and uterus.
4. Presence of submucosal and intramural fibroids larger than 5 cm or the presence of uterine polyps and congenital uterine malformations.
5. The cause of severe male infertility (TESE, PESA).

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Occyte maturity rate | 24 hours post oocyte retrieval day
  Oocyte maturity was defined as the ratio of metaphase II (MII) oocytes to the number of collected oocytes in thepatients undergoing with ICSI.

SECONDARY OUTCOMES:
Fertilization rate | 48 hours post IVF/ICSI
  Fertilization rate was defined as the ratio of normal fertilized oocytes (2PNs) to the number of oocytes used for fertilization.
Quality of obtained embryos | 48 or 72 hours after oocyte retrieval
  Embryo quality were determined according to the number of cells, the amount of fragmentation, the variation in cell size and overall symmetry (perfect, moderately asymmetric, and severely asymmetric in size and shape of the cells at Day 2 or Day 3 after oocyte retrieval:
  Excellent (Day 3: 6-8 even size blastomeres with ≤10% fragmentation), Good (Day 3: 6-8 even or uneven size blastomeres with 10%-20% fragmentation), Poor (Uneven and few blastomeres with >20% fragmentation)
Implantation rate | 1 month post embryo transfer
  The number of gestational sacs observed at trans-vaginal ultrasonography screening at 6 weeks of pregnancy divided by the number of embryos transferred.
Clinical pregnancy rate | 6-8 weeks of gestation
  Clinical pregnancy rate per transfer as defined by the presence of a gestational sac with heart beat on ultrasound at 6-8 weeks of gestation
ongoing pregnancy rate | 20 weeks after the embryos transfer
  Ongoing pregnancy was defined as a pregnancy documented by ultrasound at 20 gestational weeks that showed the presence of fetal heartbeat.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Hafezi, MD., Study Director — Department of Endocrinology and Female Infertility, Royan Institute
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- [Derived] Hafezi M, Arabipoor A, Ghaffari F, Vesali S, Zareei M, Hessari ZH. Adding L-carnitine to antagonist ovarian stimulation doesn't improve the outcomes of IVF/ ICSI cycle in patients with polycystic ovarian syndrome: a double-blind randomized clinical trial. J Ovarian Res. 2024 Jan 9;17(1):9. doi: 10.1186/s13048-023-01319-7. PMID 38191449